CLINICAL TRIAL: NCT02806791
Title: Efficacy of Biosimilar Filgrastim on the Mobilization of Hematopoietic Stem Cell CD34+ (Cluster of Differentiation 34) and on the Kinetic Engraftment After Autologous Transplant in Patients With Blood Cancers
Brief Title: Efficacy of Biosimilar Filgrastim on the Mobilization of Hematopoietic Stem Cell CD34+ (Cluster of Differentiation 34) and on the Kinetic Engraftment
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: Azienda Ospedaliera San Giovanni Battista (Other)
Responsible Party: Principal Investigator, Benedetto Bruno, Program Head, Bone Marrow Transplantation Unit, Azienda Ospedaliera San Giovanni Battista
Other Study IDs: BIO-AUTO 06-15
Record Dates: First submitted 2016-05-31; First posted 2016-06-21 (Estimated); Last update posted 2016-06-21 (Estimated); Status verified 2016-06

CONDITIONS: Blood Diseases
Keywords: Patients
MeSH Terms: conditions — Hematologic Diseases | interventions — Filgrastim

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective

INTERVENTIONS:
Drug: FILGRASTIM

SUMMARY:
The endogenous growth factor granulocyte (G-CSF) stimulates the proliferation and differentiation of hematopoietic progenitors commissioned to mature as neutrophils and activated granulocytes mature neutrophils. In the field of hematology oncology G-CSF it is used to reduce the duration and complications of chemotherapy-induced neutropenia and to stimulate the mobilization and subsequent collection of circulating hematopoietic stem cells in order to use them for autologous transplantation procedure.

Filgrastim and Lenograstim originator are marketed for many years and are considered the reference molecules for the production of biosimilar.

For several years it is available and entered into common clinical practice the use of filgrastim biosimilar (Bio-GCSF) in treating the patient oncohematologic.

Aim of the study is to analyze retrospectively a large series of patients and assess the impacts of the Bio-GCSF on the collection of hematopoietic stem cells and recovery of blood counts post autologous transplantation; the data will be compared with a historical cohort of reference that has been treated with G-CSF originator.

The study results will not generate any diagnostic or therapeutic intervention in patients still alive.

ELIGIBILITY:
Inclusion Criteria:

* > 18 years with history of autologous transplant
* hematological diseases including:
* Multiple Myeloma
* Hodgkin's Lymphoma
* Non-Hodgkin lymphoma B and T
* Lymphocytic leukemia
* Acute myeloid leukemia

Exclusion Criteria:

* N.A.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients with Blood Cancer
Sampling Method: Non-Probability Sample
Enrollment: 300 (Actual)
Dates: Start 2016-05; Primary Completion 2016-05 (Actual)

PRIMARY OUTCOMES:
Collection of autologous stem cells (time the median of achieving> 20 CD34 + / ul circulating) | until reaching 20,000 platelets (2006-2015)
Trend in blood counts after discharge values | Until day +75 post autologous transplantation (2006-2015)
Collection of autologous stem cells (total hematopoietic stem cells CD34 + * 10 ^ 6 / kg collected) | at the moment of the collection of autologous stem cells (2006-2015)
Collection of autologous stem cells (the median time from the first day of chemotherapy mobilizing) | from the first day of chemotherapy mobilizing (2006-2015)
  the median time (in days) from the first day of chemotherapy mobilizing the effective collection of stem cells
Collection of autologous stem cells (the median number of leukapheresis performed) | at the moment of the collection of autologous stem cells (2006-2015)
Collection of autologous stem cells (median number of white blood cells) | at the moment of the collection of autologous stem cells
  the median number of white blood cells in the process of mobilization
Collection of autologous stem cells ( with the aid of Plerixafor) | at the moment of the collection of autologous stem cells (2006-2015)
  the proportion of patients who have the mobilized peripheral blood stem cells with the aid of Plerixafor
Engraftment after autologous transplantation (granulocyte and platelet engraftment) | from transplant to engraftment (2006-2015)
  cumulative incidence of granulocyte and platelet engraftment
Engraftment after autologous transplantation ( median time to achieve neutrophils> 500) | from transplant to platelets engraftment (2006-2015)
  the median time to achieve neutrophils> 500 / ul for 3 consecutive days / platelets> 20,000 / ul for 7 consecutive days
Engraftment after autologous transplantation (the median number of days of G-CSF administration) | from transplant to engraftment (2006-2015)
Engraftment after autologous transplantation (median number of days of aplasia) | from transplant to engraftment (2006-2015)
Engraftment after autologous transplantation (median length of stay) | from transplant to engraftment (2006-2015)
Engraftment after autologous transplantation (number of transfusions) | from transplant to platelets engraftment (2006-2015)
  number of transfusions of packed red cells and platelet pool / patient needed

SECONDARY OUTCOMES:
transplant-related mortality | from transplant to death (if applicable) (2006-2015)
Overall survival (overall survival, OS) | to a year from autologous (2006-2015)

CONTACTS AND LOCATIONS:
Locations (1):
- Aou Citta' Della Salute E Della Scienza Di Torino, Divisione Di Ematologia, Sscvd Trapianto Allogenico, Torino, Italy